CLINICAL TRIAL: NCT00363181
Title: Does Olanzapine Inhibit the Secretory Response to Insulin Resistance?
Brief Title: Side Effects of Antipsychotic Medications
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: F1DMC-X280
Record Dates: First submitted 2006-08-09; First posted 2006-08-15 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Insulin Resistance; Metabolic Syndrome X; Schizophrenia and Disorders With Psychotic Features; Mood Disorders; Psychotic Disorders
Keywords: Insulin resistance; Metabolic problems; Weight gain; Mental health problems; Mental disorders; Antipsychotic medication; Olanzapine
MeSH Terms: conditions — Insulin Resistance; Metabolic Syndrome; Schizophrenia Spectrum and Other Psychotic Disorders; Mood Disorders; Psychotic Disorders; Weight Gain; Mental Disorders

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Medications like olanzapine have been associated with the development of weight gain and diabetes in some patients. It is not known if the increased risk of developing diabetes is a direct effect on insulin or simply related to weight gain.

We hope to learn in this study whether or not olanzapine directly slows down insulin secretion from the pancreas, thereby increasing the risk of developing diabetes.

DETAILED DESCRIPTION:
Objectives: The use of atypical antipsychotics has been associated with increased weight gain, the development of type-2 diabetes, and, in rare cases, diabetic ketoacidosis. It is not clear if these changes are a direct function of antipsychotics on either insulin action or insulin secretion, or simply related to their ability to induce weight gain in a population at increased risk to develop hyperglycemia. The objective of this investigation is to determine if treatment with the atypical antipsychotics olanzapine impairs the ability of the pancreatic beta cell to increase its insulin secretory response to graded increases in plasma glucose concentration in non-diabetic, insulin resistant individuals. In addition, we will compare the range of insulin-mediated glucose uptake (IMGU) in olanzapine-treated versus non-antipsychotic treated patients.

Research Plan and Methods: 120 subjects with psychiatric disorders will be enrolled; 60 patients on olanzapine and 60 patients with similar psychiatric diagnoses on a different antipsychotic medication (ziprasidone, risperidone or aripiprazole). All subjects will have a fasting plasma glucose concentration <126 mg/dL, and on no medication with a direct effect on IMGU. Subjects will be admitted to the General Clinical Research Center (GCRC) at Stanford Medical Center and evaluated by an insulin suppression test (IST) to determine their IMGU. Subjects with a steady state plasma glucose (SSPG) concentration during the IST that is >180 mg/dL will be defined as being insulin resistant. From this population of subjects, 15 patients on olanzapine and 15 patients not on any antipsychotic, will return to the GCRC to determine their glucose-stimulated insulin secretory dose-response curves (GS-ISR). The GS-ISR at the same glucose concentration will be compared between the subjects on olanzapine (n=15) and the not on an antipsychotic (n=15) by analysis of variance. Analyses of the 120 subjects screened for insulin resistance will compare 1) the means and distribution of the SSPG concentrations in olanzapine and non-olanzapine treated patients with psychiatric diagnoses; and 2) the means of the two experimental groups with psychiatric diagnoses to Dr. Reaven's data base of volunteers without psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* Participants 30-66 years of age
* Body mass index (BMI) >25 < 35 kg/m2.
* Fasting plasma glucose concentration < 126 mg/dL
* Stable on one of the following psychiatric medication: Olanzapine (Zyprexa®), Ziprasidone (Geodon®), Aripiprazole (Abilify®), or Risperidone (Risperdal®)
* Stable on psychiatric medication for at least 3 months

Exclusion Criteria:

* Medications that directly affect insulin-mediated glucose disposal
* Intense suicidal impulses/intent
* Alcohol or substance abuse for 3 months.
* Major medical problems, i.e., clinically unstable medical disorder or condition; cardiovascular, hepatic, renal, gastrointestinal, pulmonary, endocrine or other systemic disease that would, in the investigator's clinical judgment interfere with the endocrine measures obtained in this study.

Ages: 30 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Lindley, MD, PhD, Principal Investigator — Stanford School of Medicine / VA Palo Alto; Gerald M Reaven, MD, Principal Investigator — Stanford School of Medicine
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No